CLINICAL TRIAL: NCT00276796
Title: A Limited Access Phase II Trial of Weekly Topotecan (NSC #609699), Paclitaxel (NSC #673089), and Cisplatin (NSC #119875) in the Treatment of Advanced, Persistent, or Recurrent Carcinoma of the Cervix
Brief Title: Paclitaxel, Topotecan, and Cisplatin in Treating Patients With Advanced, Persistent, or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Philip J. DiSaia, Gynecologic Oncology Group
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456248; GOG-0076EE
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2009-02

CONDITIONS: Cervical Cancer
Keywords: cervical squamous cell carcinoma; stage III cervical cancer; recurrent cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical small cell carcinoma; stage IVA cervical cancer; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Paclitaxel; Topotecan

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, topotecan, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with topotecan and cisplatin works in treating patients with advanced, persistent, or recurrent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the antitumor activity of the combination of paclitaxel, topotecan, and cisplatin in patients with advanced, persistent, or recurrent carcinoma of the cervix.
* Determine the nature and degree of toxicity for this drug regimen in these patients.

Secondary

* Determine the duration of progression-free survival and overall survival.
* Determine the impact of prior chemoradiation on response to treatment.

OUTLINE: This is an open-label study.

Patients receive paclitaxel IV over 1 hour followed by topotecan IV over 30 minutes and cisplatin IV over 1 hour on days 1 and 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 66 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Advanced, persistent, or recurrent squamous or nonsquamous cell carcinoma of the cervix with documented disease progression

  * Histologic confirmation of the original primary tumor is required
* Disease must be measurable in at least one dimension by conventional techniques, including palpation, plain x-ray, CT scan, or MRI

  * Measurable disease is defined as at least one lesion that can be accurately measured
  * Each lesion must be ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
  * Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence ≥ 90 days after completion of radiation therapy

PATIENT CHARACTERISTICS:

* GOG performance status 0-2
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT and alkaline phosphatase ≤ 2.5 times ULN
* Neuropathy (sensory and motor) ≤ grade 1
* No active infection requiring antibiotics
* No evidence of more than one malignancy present within the past 5 years

  * Nonmelanoma skin cancer allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior therapy with cytotoxic drugs for advanced or recurrent cervical carcinoma

  * Prior cisplatin as a radiosensitizer for primary treatment of disease allowed
* No previous cancer treatment that contraindicates study treatment
* No prior radiotherapy to any portion of the abdominal cavity or pelvis except for the treatment of cervical cancer
* No prior chemotherapy for any abdominal or pelvic tumor except for the treatment of cervical cancer
* Recovered from effects of recent surgery, radiotherapy, or other therapy
* At least 4 weeks since prior radiotherapy
* More than 3 years since prior radiotherapy for localized cancer of the breast, head and neck, or skin and free of recurrent or metastatic disease
* More than 3 years since prior adjuvant chemotherapy for localized breast cancer provided patient is free of recurrent or metastatic disease
* No hormonal therapy directed at the malignant tumor within the past week
* Concurrent hormone replacement therapy is permitted
* No concurrent amifostine or other protective reagents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The frequency and duration of objective response
The frequency and severity of observed adverse effects

SECONDARY OUTCOMES:
Progression-free survival and overall survival
Prognostic factor: prior chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Harry J. Long, MD, Study Chair — Mayo Clinic